CLINICAL TRIAL: NCT06400836
Title: Impact of Carbohydrate Timing on Glucose Metabolism and Substrate Oxidation Following High-Intensity Evening Aerobic Exercise in Athletes: A Randomized Controlled Study
Brief Title: Nutrient Timing in Connection to Evening Exercise
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Göteborg University (Other)
Collaborators: Örebro University, Sweden (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: Dnr: 2022-03056-01
Record Dates: First submitted 2024-04-11; First posted 2024-05-06 (Actual); Last update posted 2024-05-06 (Actual); Status verified 2024-05

CONDITIONS: Carbohydrate Metabolism; Lipid Metabolism; Blood Glucose; Oral Glucose Tolerance Test
Keywords: Athletes; Continuous glucose monitoring; Exercise; Metabolism; Nutrition
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Intervention Model Description: Crossover Assignment Randomised double-blind cross-over study
Who Masked: Participant, Investigator
Masking Description: Double (Participant, Investigator)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Carbohydrate drink (Active Comparator): All study participants will receive the carbohydrate (CHO) drink and the placebo in a randomized, doubleblind crossover fashion. The CHO drink and placebo products have similar appearance and taste.
  Interventions: Other: Carbohydrate timing - carbohydrate intake before or after exercise
- Placebo (Placebo Comparator): All study participants will receive the carbohydrate (CHO) drink and the placebo in a randomized, double-blind crossover fashion. The CHO drink and placebo products have similar appearance and taste.
  Interventions: Other: Carbohydrate timing - carbohydrate intake before or after exercise

INTERVENTIONS:
Other: Carbohydrate timing - carbohydrate intake before or after exercise — The study aims to investigate how pre- or post evening exercise carbohydrate ingestion influences glucose metabolism and substrate oxidation (fat/CHO) during exercise and after exercise in athletes during the nocturnal period (21:00-06:00) and the morning after during an 120 minute oral glucose tolerance test (OGTT).

SUMMARY:
Physical exercise (PE) significantly influences insulin sensitivity (IS), glucose control and overall metabolic health. While PE effectively enhances IS and glucose regulation, the timing of nutrient intake, before and after exercise, plays a crucial role in modulating its effects.

The aim of this study is to evaluate how pre- or post-evening exercise carbohydrate (CHO) ingestion influences glucose metabolism and substrate oxidation (fat/CHO) during exercise and after exercise in athletes during the nocturnal period and the morning after during an oral glucose tolerance test (OGTT).

DETAILED DESCRIPTION:
The aim of this study is to evaluate how pre- or post-evening exercise carbohydrate (CHO) ingestion influences glucose metabolism and substrate oxidation (fat/CHO) during exercise and after exercise in athletes during the nocturnal period and the morning after during an oral glucose tolerance test (OGTT).

The primary objective is to assess glucose regulation during a 120-minute OGTT the following day.

The secondary objective is to investigate substrate metabolism (CHO and fat oxidation) during a 120-minute OGTT the following day.

Ten healthy, well-trained male endurance cyclists/triathletes, aged 19-45 years, are recruited via local contacts from the Gothenburg region, Sweden. The study is performed in accordance with the Declaration of Helsinki 2008 and is approved by the Swedish Ethical Review Authority (Dnr: 2022-03056-01). All participants gave their written informed consent before inclusion.

The study has a double-blind, randomized, placebo-controlled, crossover design.

After baseline assessment and determination of maximal oxygen uptake (VO2 max), participants undergo a familiarization cycle exercise trial. This trial serves a dual purpose: first, to establish the appropriate amount of CHO to be incorporated into the pre- or post-drink for subsequent cycle experimental trials, and second, to familiarize participants with the equipment and study protocol.

Three days prior to the cycle experimental trial, subcutaneous insertion of a glucose sensor for continuous glucose monitoring (CGM) takes place. Participants are randomly assigned to consume either a CHO drink or a placebo (PLA) drink (containing no energy) two hours prior to the cycle experimental trial that starts at 19:30. During the exercise trial, participants engage in submaximal cycling exercise at 70% of their maximal workload (Wmax), followed by a 25-minute time trial (TT). The total duration of the exercise session is approximately 90 minutes. Workload during the TT is individualized based on each participant's maximal work capacity (Wmax). During exercise, capillary glucose levels, heart rate, and rate of perceived exertion (RPE; Borg category scale 6-20) are measured. Additionally, respiratory gases are collected during 5-minute periods at every 15-minute interval to assess substrate utilization.

Immediately after completing the TT, participants switch to the opposite drink condition: those who initially received the CHO drink consume the PLA drink, and vice versa. The amount of CHO in the CHO drink consumed by each participant is precisely matched to the amount of CHO that the participant oxidizes during the exercise trial.

After the ingestion of the CHO- or placebo drink, participants fast overnight. CGM technology is used to measure interstitial glucose values during the night.

At 08:00, participants consume a 300mL solution containing 75g glucose for a 120-min OGTT. Capillary blood samples are collected at baseline and every 15 minutes during the OGTT. Respiratory gases are collected to measure substrate oxidation. The same protocol is reproduced the following week, with the reverse order of the test drink intake.

Three days preceding both control and experimental trials, participants are provided with a standardized diet consisting of pre-packaged meals that match their daily energy and macronutrient needs to prevent energy deficiency.

ELIGIBILITY:
Inclusion Criteria:

* Females and males
* 18-50 years
* Endurance fitness level of ≥40 mL O2/kg/min.
* Signed informed consent

Exclusion Criteria:

• Medical treatment and/or nutritional supplements that may affect glucose tolerance, substrate oxidation and performance capacity

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2022-01-10 (Actual); Primary Completion 2022-09-02 (Actual); Study Completion 2022-09-02 (Actual)

PRIMARY OUTCOMES:
To investigate change in glucose tolerance during a 75g glucose, 120 min oral glucose tolerance test (OGTT) | Comparing the change in glucose tolerance during the OGTT between baseline (no exercise) week 0, compared to interventions week 1 and week 2 involving previous evening exercise, with carbohydrates consumed either before or after exercise.
  To quantify participants' glucose tolerance, the change in plasma glucose levels (mmol/L) will be measured over a 120-minute period following the ingestion of a standardized 75g glucose solution during an OGTT.

SECONDARY OUTCOMES:
To investigate substrate oxidation during the oral glucose tolerance test (OGTT) | Comparing the change in substrate oxidation during the OGTT between baseline (no exercise) week 0, compared to interventions week 1 and week 2 involving previous evening exercise with carbohydrates being consumed either before or after exercise.
  To quantify substrate oxidation rates (carbohydrate oxidation (g/minute) and fat oxidation (g/minute), the change in respiratory exchange ratios (RER) will be measured during the 120-minute OGTT period.

OTHER OUTCOMES:
To investigate performance capacity during a cycle ergometer time trial (TT). | Comparing the change in performance capacity between the interventions involving carbohydrates being consumed either before (week 1) or after the time trial (week 2). Note that respective arm will be randomized.
  Performance capacity was assessed by measuring the time (seconds) required to complete a specific amount of work.
To investigate substrate oxidation during 50 min submaximal evening exercise. | Comparing the change in substrate oxidation between the interventions involving previous evening exercise with carbohydrates being consumed either before (week 1) or after exercise (week 2). Note that respective arm will be randomized.
  To quantify substrate oxidation rates (carbohydrate oxidation (g/minute) and fat oxidation (g/minute), the change in respiratory exchange ratios will be measured during the 50 min submaximal exercise.
To investigate nocturnal glucose regulation. | Comparing the change in glucose levels (mmol/L) during the period 21:00-06:00 between baseline (no exercise) week 0, compared to interventions week 1 and week 2 involving previous evening exercise, with CHO consumed either before or after exercise.
  To quantify participants' nocturnal glucose regulation, the change in interstitial glucose levels (mmol/L) will be measured during the period 21:00-06:00 utilizing continuous glucose monitoring (CGM).

CONTACTS AND LOCATIONS:
Overall Officials: Stefan Pettersson, Assoc. Prof., Principal Investigator — Department of Food and Nutrition, and Sport Science, University of Gothenburg, Sweden
Locations (1):
- Department of Food and Nutrition, and Sport Science, Centre for Health and Performance, University of Gothenburg, Gothenburg, Sweden, Gothenburg, Bohuslän, Sweden

IPD SHARING:
Plan to Share IPD: No